CLINICAL TRIAL: NCT06614933
Title: How Does the Type of Waveform Affect Tolerability With Transcutaneous Auricular Vagus Nerve Stimulation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Marlon Wong, Clinical Associate Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 20240796
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be blinded to which protocol they are receiving during data collection. The investigator responsible for processing HRV data will be blinded to group assignment, and investigators will be blinded to group assignment when conducting qualitative data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Biphasic followed by monophasic taVNS group (Experimental): Participants in the group "Biphasic followed by monophasic taVNS" will be in this group for up to 6 hours.
  Interventions: Device: Biphasic transcutaneous auricular vagus nerve stimulation; Device: Monophasic transcutaneous auricular vagus nerve stimulation
- Monophasic followed by biphasic taVNS group (Active Comparator): Participants in the group "monophasic followed by biphasic" will be in this group for up to 6 hours.
  Interventions: Device: Biphasic transcutaneous auricular vagus nerve stimulation; Device: Monophasic transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: Biphasic transcutaneous auricular vagus nerve stimulation — Transauricular vagus nerve stimulation (taVNS) is a simple technique in which small surface electrodes are placed over the skin of the ear that are thought to be innervated by the auricular branch of the vagus nerve (ABVN). Participants in this group will first receive taVNS with a biphasic current, continuous at 25 Hz, for 1 hour, in-person.
Device: Monophasic transcutaneous auricular vagus nerve stimulation — Transauricular vagus nerve stimulation (taVNS) is a simple technique in which small surface electrodes are placed over the skin of the ear that are thought to be innervated by the auricular branch of the vagus nerve (ABVN). Participants in this group will first receive taVNS with a monophasic current, with a 50% duty cycle at 25 Hz, for 1-hour, in-person.

SUMMARY:
The purpose of this research study is to investigate the effects of different forms of a gentle form of electrical stimulation applied to the ear, known as transcutaneous auricular vagus nerve stimulation (taVNS). The research team is interested in how the different forms affect comfort and tolerability, as well as how well it works.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18-80 years
2. English speaking (must be able to consent and complete the interviews in English)

Exclusion Criteria:

1. chronic pain (average intensity >2/10 on 0-10 scale, for longer than 3 months)
2. acute pain of intensity greater than 3/10
3. chronic inflammatory conditions that are poorly controlled (e.g., diabetes, autoimmune disease)
4. any unstable medical condition or medical contraindication to moderate physical exertion (e.g., unstable angina or cardiac arrythmia)
5. pregnancy
6. currently taking Buprenorphine or recently stopped taking (within 1 month)
7. presence of cognitive impairment or language barrier that impairs full autonomy in the consent process or in the ability to participate in detailed interviews
8. implants in the head or neck, cochlear implants, or pacemaker
9. head or neck metastasis or recent ear trauma
10. history of epilepsy
11. history of autonomic nervous system dysfunction (e.g., postural orthostatic tachycardia syndrome).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Tolerability measured by tolerability questionnaire | Up to 3 hours.
  Tolerability will be assessed with a questionnaire with scores ranging from 0 (no discomfort)-10 (worst pain imaginable) for comfort.
Tolerability measured by self-report | Up to 3 hours.
  Tolerability will be assessed using semi-structured interviews. Investigators will ask about the sensations experienced and preferences. Participants will self-report their responses.

SECONDARY OUTCOMES:
Change in heart rate variability (HRV) | Baseline and up to 3 hours.
  HRV will be measured with an H10 chest strap device. Values after stimulation will be subtracted from baseline values; thus, a positive number will indicate an increase in HRV post taVNS.

CONTACTS AND LOCATIONS:
Overall Officials: Marlon Wong, PT, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Plumer Building, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No